CLINICAL TRIAL: NCT04568980
Title: Assessment of Contraceptive Safety and Effectiveness in Cystic Fibrosis: A Retrospective Analysis
Brief Title: Assessment of Contraceptive Safety and Effectiveness in Cystic Fibrosis
Acronym: CASE4CF
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Emily Godfrey, Associate Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00008095
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Cystic Fibrosis; Contraception
Keywords: birth control; contraception; cystic fibrosis; bone mineral density; CFTR modulator; women
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hormonal contraceptive users: Persons exposed to any hormonal method of birth control. This includes combined oral contraceptive pills, combined transdermal patch, combined vaginal ring, progestin-only pills, depo-medroxyacetate, levonorgestrel intrauterine system/device, hormonal subdermal implant
- Non-hormonal contraceptive users: Persons exposed to any non-hormonal method of birth control. This includes male or female sterilization methods, Copper intrauterine device, internal/external condoms, diaphragm, cervical cap, withdrawal, sponge, fertility based methods, spermicide
- Non-contraceptive users: Persons who did not use any method of birth control

SUMMARY:
The long-term goal is to study the safety and effectiveness of hormonal contraception for women with cystic fibrosis (CF) and contribute to national guidelines that the Cystic Fibrosis Foundation and the Centers for Disease Control and Prevention (CDC) provide to clinicians. The study objectives are to determine whether hormonal contraceptive methods improve overall pulmonary health, worsen CF-related disease or CF liver disease, or are effective against unwanted pregnancy with concomitant CF transmembrane conductance regulator (CFTR) modulator use. The hypothesis is that hormonal contraceptive methods are safe and do not worsen CF-related complications over time,improve FEV-1 when compared to non-hormonal users, and oral birth control methods with CFTR modulator use.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional, observational cohort design among reproductive-aged women (ages 18-45 years) with CF. The investigators intend to ask about 625 female participants to provide information about their types of past contraceptive use from 2008 through the most recent data available from CFFPR (2018 or 2019). Before initiating our trial among up to 625 respondents, the investigators intend to pre-test the survey questions on our self-respondent questionnaire among as many as 50 women with and without CF through CFF Community Voice, the Cystic Fibrosis Research, Inc. (CFRI), and the Cystic Fibrosis Reproductive and Sexual Health Collaborative (CFReSHC). Pre-testing the study survey questions will help ensure contraceptive, pregnancy, and other reproductive health data from respondents for the larger phase of this study are as complete and accurate as possible. Once the survey has been piloted and revised accordingly, the investigators will collect past contraceptive, pregnancy and other reproductive health data from up to 625 women at 10 different CF centers. The investigators may over-sample by 25 participants because it is possible that some participants from UW, UTSW and National Jewish may have participated an earlier published study related to contraceptive use and CFFPR. Recruiting through the CF centers will help ensure that women with a confirmed diagnosis of CF respond to the finalized survey. The investigators will link respondent self-reported contraceptive and reproductive health data with CFFPR clinical data. The investigators will ask for EMR data from the 10 different CF centers to validate DXA scan results with findings regarding osteoporosis, osteopenia, and bone fracture in the CFFPR. The investigators plan to randomly select about 10 consented subjects from each of the centers for the EMR DXA scan chart review. Because of the need to link questionnaires and clinical case report forms correctly to the same women with CF in the CFFPR clinical data, this study requests identifiable information, including the CFFPR member ID number.

ELIGIBILITY:
Inclusion Criteria:

* Women with cystic fibrosis age 18-45 years
* Enrolled as a participant of the Cystic Fibrosis Foundation Patient Registry
* Working email address
* Can read written English

Exclusion Criteria:

* History of organ transplant
* Does not have a phone number or email address in their record
* <18 years or >45 years at enrollment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with cystic fibrosis who have not used any form of contraception, or who have used contraception for protection against pregnancy or for treatment of dysmenorrhea, pelvic pain, abnormally heavy or prolonged menstrual bleeding, endometriosis, acne or amenorrhea.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary exacerbations | 2010-2018
  Annual pulmonary exacerbation rate (PEx) (defined as episodes requiring intravenous antibiotic use at home or in hospital)

SECONDARY OUTCOMES:
Lung function | 2010-2018
  Absolute change in FEV1 (in liters) measurements over time.
Thromboembolism | 2010-2018
  Incidence of venous or arterial thromboembolism. Noted on self-respondent survey (defined as blood clot requiring anticoagulation treatment)
Liver dysfunction | 2010-2018
  Incidence of gallstones requiring surgery, hepatic steatosis, hepatic cirrhosis and/or increased liver enzyme test values (ALT/GGT)
Serum glucose trends | 2010-2018
  Incidence of insulin resistance or time to CF-related diabetes requiring insulin treatment
Nutritional status | 2010-2018
  BMI trends
Bone health | 2013-2018
  DXA scan determination of osteopenia or osteoporosis
Unintended pregnancy | 2010-2018
  Absolute number of self-reported unplanned pregnancies. We will also correlate date of reported unplanned pregnancy with dates of taking a CFTR modulator
Pseudomonas aeruginosa | 2010-2018
  Rate of conversion from non-mucoid to mucoid P. aeruginosa

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Godfrey, MD, MPH, Principal Investigator — University of Washington
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital/Harvard, Boston, Massachusetts
  - Mount Sinai Beth Israel, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04568980/Prot_SAP_000.pdf